CLINICAL TRIAL: NCT06901726
Title: An Open, Randomized, Single Dose (32mg), Two-way Crossover Study on Pharmacokinetics, Pharmacodynamics, Relative Biopotency and Bioavailability of Human Insulin Enteric Coated Capsules in Healthy Chinese Male Subjects
Brief Title: Open, Randomized Crossover Study on PK, PD, Biopotency, and Bioavailability of Insulin Capsules in Healthy Chinese Males
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, PHD, MD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORA-H-CN-008
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: two-way crossover
Masking Description: This study was open for subjects, sponsor and investigators except for analytical laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human insulin enteric coated capsules in dose 32mg (Experimental): Single oral administration of human insulin enteric coated capsules in dose 32mg.
  Interventions: Drug: Human insulin enteric coated capsules in dose 32mg
- Human Insulin Injection in dose 5 IU (Active Comparator): Single subcutaneous administration of Human Insulin Injection in dose 5IU.
  Interventions: Drug: Human Insulin Injection in dose 5IU

INTERVENTIONS:
Drug: Human insulin enteric coated capsules in dose 32mg — Single oral administration of human insulin enteric coated capsules in dose 32mg (16 mg per capsule, two capsules).
  Arms: Human insulin enteric coated capsules in dose 32mg
Drug: Human Insulin Injection in dose 5IU — Single subcutaneous administration of Human Insulin Injection in dose 5IU.
  Arms: Human Insulin Injection in dose 5 IU

SUMMARY:
Pharmacokinetics and pharmacodynamics study of 2 formulations (human insulin enteric coated capsules 32mg vs. human insulin injection 5IU) Relative biopotency and bioavailability of human insulin enteric coated capsules 32mg vs. human insulin injection 5IU

DETAILED DESCRIPTION:
An open, randomized, single dose, two-way crossover study on Pharmacokinetics, pharmacodynamics, relative biopotency and bioavailability of human insulin enteric coated capsules in healthy Chinese male subjects using hyperinsulinemic-euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male subjects aged 20-35 (inclusive);
2. Body mass index (BMI) between 19 and 24 kg/m2 ( extrems inclusive, body mass index= body weight/ height2);
3. Normal oral glucose tolerance Test (fasting plasma glucose [FPG]< 6.1 mmol/L and 2-hour postprandial blood glucose after loading with glucose [2hPG]< 7.8 mmol/L), and HbA1C<6.0%
4. Normal insulin releasing test (judged by investigator);
5. Considered generally healthy upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, without history of acute and chronic diseases with clinical significance, incl.: of the cardiovascular system, bronchopulmonary, neuroendocrine systems, endocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood, as judged by the Investigator.
6. Signed informed consent and volunteers' consent to all restrictions imposed during the study.

Exclusion Criteria:

1. Known allergic or suspected hypersensitivity to investigational product (IP) or related product
2. Previous or existing diseases of the cardiovascular system, endocrine system, gastrointestinal system, nervous system, or diseases of the lungs, hematologic, immunology, psychiatry, and metabolic abnormalities, as judged by the investigator;
3. History of heavy smoking, alcohol abuse, and drug abuse;
4. Taking more than 14 units alcohol per week within 3 months prior to screening (1unit≈360 mL of beer, 45mL of spirits, or 150 mL of wine), or receiving alcohol within 48 hours prior to IP administration, or failure to abstain from alcohol during the trial;
5. Receiving excessive amounts of tea, coffee, and/or caffeine rich beverages (8 or more cups, 1 cup ≈ 250 mL) per day within 3 months prior to screening;
6. Use of any medication that may affect glucose lowering effect (such as oral contraceptives, corticosteroids, diuretics, adrenaline, salbutamol, glucagon, growth hormone, thyroid hormone, etc.) within 28 days prior to screening;
7. Taking any medications, vitamin products, or any Chinese herbal medicine or nutrition supplements within 2 weeks prior to IP administration;
8. Participation in any clinical trial less than 3 months prior to screening or planning to participate in other trials after ICF signed.
9. Blood donation or blood loss≥ 200mL of any reasons within 3 months prior to screening; history of blood transfusion or component blood transfusion; failure to guarantee not to donate whole blood / component blood (such as plasma, platelets) during the trial or within 30 days after the end of the trial;
10. Undergo surgery prior to IP administration within 1month or plan to undergo surgery during the trial;
11. Occurrence of acute disease during screening;
12. Positive test of any: HIV-Ab, HBSAg, HCV-Ab,TP-Ab;
13. History of needle phobia and blood phobia;
14. Any conditions that make volunteer participation ineligible judged by investigating physician.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
GIRmax | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PD endpoint: The maximum glucose infusion rate
TGIRmax | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PD endpoint: The time to maximum observed glucose infusion rate
AUCGIR 0-11h | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PD endpoint: The area under the glucose infusion rate curve from 0 to 11 hours
AUCGIR0-∞ | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PD endpoint: The area under the glucose infusion rate curve from 0 to infinity

SECONDARY OUTCOMES:
Cmax | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PK endpoint: The maximum observed insulin concentration
Tmax | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PK endpoint: The time to maximum observed insulin concentration
AUCIns0-11h | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PK endpoint: The area under the insulin concentration curve from 0 to 11 hours
AUCIns0-∞ | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  PK endpoint: The area under the insulin concentration-time curve from 0 hours to infinity

OTHER OUTCOMES:
Relative biopotency | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  (AUCGIR of capsule:dosage)/(AUCGIR of injection:dosage)
Relative bioavailability | 0-11 hours (hyperinsulinemic-euglycemic clamp)
  (AUCins of capsule:dosage)/(AUCins of injection:dosage)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to Day 14
  Number of participants experiencing treatment-emergent adverse events